CLINICAL TRIAL: NCT01799616
Title: Efficiency and Safety Study of Pamidronate in Inflammatory Back Pain Due to Degenerative Disk Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: INSERM CIC 501 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0148; 2012-003569-16
Record Dates: First submitted 2013-02-21; First posted 2013-02-27 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Intervertebral Disc Degeneration; Modic I Discopathy; Back Pain; Low Back Pain; Magnetic Resonance Imaging (MRI)
Keywords: MODIC changes; Chronic low back pain; Pamidronate; Magnetic resonance imaging; Vertebrae; Intervertebral disc
MeSH Terms: conditions — Intervertebral Disc Degeneration; Back Pain; Low Back Pain | interventions — Pamidronate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Pamidronate (Experimental): In total, 48 patients will need to be recruited. These patients will be randomly assigned to one of the two groups, with each group comprising 24 patients: one group will be given pamidronate and the other placebo
  Interventions: Drug: Pamidronate
- Placebo (Other): In total, 48 patients will need to be recruited. These patients will be randomly assigned to one of the two groups, with each group comprising 24 patients: one group will be given pamidronate and the other placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pamidronate
  Arms: Pamidronate
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether pamidronate is effective and well-tolerated in the treatment of painful degenerative disk disease, also known as Modic type 1 changes

DETAILED DESCRIPTION:
Erosive degenerative disk disease, also known as Modic type 1 changes, is usually characterized by low back pain, with an inflammatory pain pattern, as seen in spondylarthropathies. Intravenous pamidronate has proven effective in patients with ankylosing spondylitis, and in painful bone diseases in general. We therefore hypothesized that pamidronate would be effective in treating back pain associated with Modic type 1 changes.

This study aimed to determine pamidronate's efficiency in reducing pain, with the primary outcome being a between-group difference of 30 points on a 100mm VAS at 3 months. Secondary outcomes are the improvement in functional status and the drug's tolerance. Primary and secondary outcome criteria will be assessed at each visit (inclusion, at 6 weeks, 3 months, and 6 months). If the primary goal is not attained, a rigid or semi-rigid back brace will be proposed to the patient, regardless of the treatment group.

In total, 48 patients will need to be recruited. These patients will be randomly assigned to one of the two groups, with each group comprising 24 patients: one group will be given pamidronate and the other placebo. Pamidronate will be administered at a dose of 90mg per day, 2 days in a row, and every patient, regardless of the treatment group, will be given paracetamol, in order to maintain blinding by preventing drug-induced fever.

ELIGIBILITY:
Inclusion Criteria:

* - Age from 18 to 60 years old
* Low back pain
* Daily pain since at least 3 months
* VAS for pain > 40/100 during the last 48 hours
* Inefficiency, intolerance, or contraindication to NSAIDS
* Inefficiency of a rigid or half-rigid back brace
* Modic 1 discopathy (diagnosed on MRI and confirmed by trained radiologist)
* Dental check-up within the last 6 months
* Signed informed consent

Exclusion Criteria:

* - Static disorders of the spine
* Contraindication to pamidronate (hypocalcemia, severe kidney failure, or allergy)
* Underage patients, patients under the protection of the law
* Previous treatment with bisphosphonates
* Pregnancy
* Local or general infection
* Previous discal surgery
* Systemic corticosteroid therapy in the last month
* Epidural or facet joint corticosteroid injection in the last month
* History of septic spondylodiscitis
* Ankylosing spondylitis
* Low back pain associated with radiculalgia
* Active psychiatric disorder
* Inability to read or understand French
* Body temperature above 38°C (fever) or Erythrocyte Sedimentation Rate above 20mm/hour

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
back pain assessed on a100mm VAS | at 3 months

SECONDARY OUTCOMES:
- Functional status using EIFEL, Dallas, FABQ, MacTar, and MCII/PASS questionnaires | at 6 weeks, 3 months, and 6 months
Back stiffness assessed by Schober's test and finger-to-floor distance | at 6 weeks, 3 months, and 6 months
Inflammatory pain pattern | at 6 weeks, 3 months, and 6 months
  Inflammatory pain pattern: number of nightly awakenings, as well as duration and intensity of morning stiffness on a 100mm VAS
assess the efficacy of a rigid back brace in treating back pain | at 6 weeks, 3 months, and 6 months
  In case of failure to reduce the pain with pamidronate at 3 months: assess the efficacy of a rigid back brace in treating back pain
Tolerance based on the number and types of side-effects | at 6 weeks, 3 months, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin SOUBRIER, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Cecchetti S, Pereira B, Roche A, Deschaumes C, Abdi D, Coudeyre E, Dubost JJ, Mathieu S, Malochet-Guinamand S, Tournadre A, Couderc M, Vayssade M, Daron C, Soubrier M. Efficacy and safety of pamidronate in Modic type 1 changes: study protocol for a prospective randomized controlled clinical trial. Trials. 2014 Apr 9;15:117. doi: 10.1186/1745-6215-15-117. PMID 24716739